CLINICAL TRIAL: NCT02476136
Title: Initial Severity and Antidepressant Efficacy for Anxiety Disorders: an Individual Patient Data Meta-analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: prof. Peter de Jonge (Other)
Responsible Party: Sponsor-Investigator, prof. Peter de Jonge, Professor of Psychiatric Epidemiology, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Other Study IDs: CSDR-1173
Record Dates: First submitted 2015-06-03; First posted 2015-06-19 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Anxiety Disorders; Panic Disorder; Obsessive-compulsive Disorder; Post-traumatic Stress Disorder; Generalized Anxiety Disorder; Social Anxiety Disorder
Keywords: individual patient data meta-analysis; anxiety disorder; antidepressants; selective serotonin reuptake inhibitors; serotonin-norepinephrine reuptake inhibitors
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic; Generalized Anxiety Disorder; Phobia, Social | interventions — Paroxetine; Duloxetine Hydrochloride; Fluoxetine; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Placebo group: Patients participating in one of the included randomized controlled trials, assigned to the placebo group
- Intervention group: Patients participating in one of the included randomized controlled trials, assigned to the investigational antidepressant (paroxetine, duloxetine or fluoxetine) or active comparator (venlafaxine) group.
  Interventions: Drug: paroxetine, duloxetine, fluoxetine or venlafaxine

INTERVENTIONS:
Drug: paroxetine, duloxetine, fluoxetine or venlafaxine
  Other Names: Paxil; Cymbalta; Prozac; Effexor
  Groups: Intervention group

SUMMARY:
Anxiety disorders are common disorders, which pose a major burden to society and the individual. An anxiety disorder may be treated with medication, in particular with antidepressants such as the selective serotonin reuptake inhibitors (SSRIs). However, much of what is known about antidepressants is derived from research in depression rather than anxiety. In recent years, researchers have found that antidepressants are more effective for severely depressed patients than they are for patients with milder symptoms. It is possible that a similar relationship between symptom severity and antidepressant efficacy exists for anxiety disorders, but there is currently little evidence available to answer this question. As antidepressants are frequently prescribed to patients with mild or moderate anxiety, a clear understanding of their effectiveness across the severity range is vital to inform treatment decisions. Therefore, the purpose of this meta-analysis is to examine whether initial symptom severity affects antidepressant efficacy for anxiety disorders.

DETAILED DESCRIPTION:
Study design:

The proposed project is an individual patient data meta-analysis. The investigators will collate data from 29 randomized controlled trials of second-generation antidepressants (specifically: paroxetine, paroxetine controlled release (CR), duloxetine, and fluoxetine) for the short-term treatment of an anxiety disorder, including a total of approximately 8,800 participants. The anxiety disorders that are included in the proposed project are generalized anxiety disorder (GAD), social anxiety disorder (SAD), obsessive-compulsive disorder (OCD), post-traumatic stress disorder (PTSD), and panic disorder (PD). Generalized linear mixed models will be used to investigate whether initial symptom severity is related to antidepressant efficacy.

Statistical analysis plan:

A separate longitudinal analysis will be conducted for each disorder. For GAD, SAD, OCD, and PTSD, linear mixed models will be used; for PD, a generalized linear mixed model (multilevel negative binomial regression) will be used, as the dependent variable for this disorder (number of panic attacks) is a discrete count variable. Maximum likelihood estimation will be used as the estimation method for the linear mixed models, while Laplace approximation will be used as the estimation method for the multilevel negative binomial regression for PD. In all models, measurement occasion represents level 1, participants represent level 2, and trial represents level 3. The effect measure of interest is the change in symptoms from baseline, except for PD, for which the effect measure of interest is the total number of panic attacks per two weeks.

The initial model will be built by including all the fixed effects of interest, regardless of significance. These include initial severity, treatment group and covariates (see below). Linear and quadratic terms for time (in days since baseline) will be included. For each participant, the actual visit dates will be used (if available) rather than the intended weekly visit date. The following two- and three-way interactions will also be included: severity x group, severity x linear time, group x linear time, severity x group x linear time, severity x quadratic time, group x quadratic time, severity x group x quadratic time.

Using this first model, the variance-covariance structure of the nested data will be modeled by including random effects. Random effects for study, subject and (linear and quadratic) time, as well as various covariance structures (unstructured, autocorrelated errors, Toeplitz, etc.) will be considered. Restricted maximum likelihood (REML) will be used for estimation, and the best-fitting model will be selected based upon the Akaike Information Criterion (AICc).

In this best-fitting model, backward selection with maximum likelihood (ML) will be used to select the significant fixed effects. Non-significant interaction terms will be removed from the model (unless the three-way interaction of group x severity x (linear or quadratic) time is significant, in which case all two-way interactions and main effects that use these variables will be retained). The best-fitting model will again be selected based upon the Akaike Information Criterion (AICc).

Covariates: Models with and without the following covariates will be tested: age, gender, and duration of illness (if available). Only the main effect of these covariates will be included; no interactions with other variables will be included.

Missing data: Baseline variables (such as initial severity) are likely to be essentially complete, but some change scores are likely to be missing due to dropout or missed measurement occasions. The assumption is made that these data are missing at random (MAR), that is: missingness of the dependent variable may depend upon observed variables (such as previous symptom scores or covariates), but it does not depend upon the value of the unobserved (missing) variable. When MAR holds, the mixed model yields unbiased estimates of coefficients and standard errors even when some data is missing, and no other methods for handling missing data are required.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in the intent-to-treat population of a randomized controlled trial of a second-generation antidepressant for the short-term treatment of an anxiety disorder
* Diagnosed with an anxiety disorder (GAD, SAD, OCD, PTSD or PD)

Exclusion Criteria:

* Assignment to an active comparator that is not a second-generation antidepressant (e.g. a benzodiazepine)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of adults aged 18 and older (with the exception of OCD trials, which may include adolescents aged 14 and older) who have been diagnosed with generalized anxiety disorder (GAD), social anxiety disorder (SAD), obsessive-compulsive disorder (OCD), post-traumatic stress disorder (PTSD), or panic disorder (PD) and who were randomized to placebo or to treatment with a second-generation antidepressant.
Sampling Method: Non-Probability Sample
Enrollment: 8800 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the Hamilton Anxiety Rating Scale (HAM-A) | Baseline to trial endpoint (8 to 10 weeks)
Change from baseline on the Liebowitz Social Anxiety Scale (LSAS) | Baseline to trial endpoint (12 weeks)
Change from baseline on the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) | Baseline to trial endpoint (12 to 13 weeks)
Change from baseline on the Clinician-Administered PTSD Scale (CAPS) | Baseline to trial endpoint (12 weeks)
The total number of panic attacks | Baseline to trial endpoint (10 to 12 weeks)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vries YA, Roest AM, Burgerhof JGM, de Jonge P. Initial severity and antidepressant efficacy for anxiety disorders, obsessive-compulsive disorder, and posttraumatic stress disorder: An individual patient data meta-analysis. Depress Anxiety. 2018 Jun;35(6):515-522. doi: 10.1002/da.22737. Epub 2018 Apr 16. PMID 29659102